CLINICAL TRIAL: NCT05932264
Title: A Phase II Study of Efficacy and Safety of Combination of Apatinib and Fluzoparib With or Without Adebrelimab in Previously-treated TP53-mutant Advanced Non-small Cell Lung Cancer
Brief Title: Apatinib and Fluzoparib With or Without Adebrelimab in Previously-treated TP53-mutant Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2023-205-01/MA-NSCLC-II-029
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: NSCLC; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib; fluzoparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Apatinib + Fluzoparib (Experimental)
  Interventions: Drug: Apatinib + Fluzoparib
- Cohort 2: Apatinib + Fluzoparib + Adebrelimab (Experimental)
  Interventions: Drug: Apatinib + Fluzoparib + Adebrelimab

INTERVENTIONS:
Drug: Apatinib + Fluzoparib — Cohort 1: Apatinib 375 mg po qd; Fluzoparib 100mg po bid
  Arms: Cohort 1: Apatinib + Fluzoparib
Drug: Apatinib + Fluzoparib + Adebrelimab — Cohort 2: Apatinib 375 mg po qd; Fluzoparib 100mg po bid; Adebrelimab 1200mg, iv, d1, q3w]
  Arms: Cohort 2: Apatinib + Fluzoparib + Adebrelimab

SUMMARY:
This is a phase 2, open-label study to evaluate the efficacy and safety of combination of Apatinib and Fluzoparib with or without Adebrelimab in previously-treated TP53-mutant advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This study is an open-label, prospective phase II study to evaluate the efficacy and safety of of combination of Apatinib and Fluzoparib with or without Adebrelimab in previously-treated TP53-mutant advanced non-small cell lung cancer. The study is divided into 2 cohorts. Cohort 1 is a two-drug cohort [Apatinib 375 mg po qd; Fluzoparib 100mg po bid], and cohort 2 is a three-drug cohort [apatinib 375 mg po qd; fluzoparib 100mg po bid; Adebrelimab 1200mg, iv, d1, q3w]. The sample sizes of these two cohorts were determined according to Simon's Two-Stage Design, and enrollment of cohort 2 will be initiated after the enrollment of cohort 1 is completed. Ultimately, 34 patients are enrolled in the cohort 1 and 26 in the cohort 2.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate and sign the informed consent in person
2. Male or female patients, aged ≥18 years and ≤75 years
3. Histologically or cytologically confirmed non-small cell lung cancer with clinical stage IIIB-IV (International Association for the Study of Lung Cancer, 8th Edition)
4. TP53 gain-of-function mutations (P151S, Y163C, R175H, L194R, Y220C, R248Q, R248W, R249S, R273C, R273H, R273L, R151S, Y163C, R175H, L194R, R220C, R248W, R249S, R273C, R273H, R273L, R282W) or p53 protein high expression (≥80% nuclear staining positive) confirmed by immunohistochemistry; Consent to provide previously stored tumor tissue specimens or fresh biopsy tumor lesion tissue
5. Have at least one measurable lesion (RECIST 1.1 criteria)
6. Disease has been progressed after the approved first-line therapy. In brief, patients with positive driver genes (EGFR, ALK, ROS1, BRAF, MET, RET) must have received the corresponding targeted therapy approved in China, and were subsequently treated with platinum-based standard chemotherapy; Patients who are negative for driver genes have to be previously treated with approved chemoimmunotherapy.
7. ECOG score 0-1
8. Expected survival time ≥12 weeks, as assessed by the investigator.
9. Normal organ function, includes:

   1. Neutrophil count ≥1.5 × 10^9 / L,
   2. Platelet count ≥100 × 10^9 / L,
   3. Hemoglobin ≥10 g/dL
   4. Serum creatinine ≤1.5× upper limit of normal (ULN), creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula)
   5. Total bilirubin ≤ 1.5×ULN
   6. AST and ALT ≤ 2.5×ULN; Patients with liver metastasis, AST and ALT≤5×ULN, were determined by the investigator
   7. Normal coagulation function: INR and PT≤ 1.5 ×ULN
10. The pregnancy test is negative at enrollment. To be enrolled, men or women are required to commit to using adequate, effective contraception or abstinence from sex from the start of the study until the end of the study and for 3 months after the last dose of the study drug
11. The toxic effects of any previous treatment have returned to ≤CTCAE1 or baseline level
12. Stopping other antineoplastic therapy including but not limited to chemotherapy, radiotherapy and surgery 4 weeks before receiving the study drugs; targeted therapy should be discontinued for at least 5 half-lives of the corresponding drug before receiving the study drugs.

Exclusion Criteria:

1. Non-small cell lung cancer admixed with components of small cell lung cancer or sarcomatoid carcinoma, as confirmed by histology or cytology.
2. Patients with > 2 lines of prior chemotherapy, or previously treated with PARP inhibitor or small-molecule angiogenesis inhibitors.
3. Patients with coagulation disorders or who are considered to have a risk of hemorrhage, or the tumor had invades the large blood vessels or wrapped the blood vessels with unclear boundaries on CT or MR imaging.
4. Patients with a known allergy to the active or inactive ingredient of any of the drugs in the study, or a history of severe hypersensitivity reaction to any monoclonal antibody
5. Symptomatic, uncontrolled brain or leptomeningeal metastases
6. Had undergone major surgery within 4 weeks before the start of the study, or had complications/sequelae that have not yet recovered
7. Patients with previously or currently diagnosed myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
8. Suffering from serious or uncontrolled illness, including but not limited to:

   Uncontrollable nausea and vomiting, intestinal obstruction, inability to swallow the study drug, and any gastrointestinal disorders that may interfere with the absorption and metabolism of the drug.
9. Patients with respiratory syndrome due to pleural effusion or ascites (≥CTCAE grade 2 dyspnea)
10. Active viral infections such as human immunodeficiency virus, hepatitis B, hepatitis C, etc
11. Uncontrolled grand mal seizures, unstable spinal cord compression, superior vena cava syndrome, or other mental disorders that prevent the patient from signing informed consent
12. Immunodeficiency (other than splenectomy), or other conditions considered by the investigator to be likely to expose the patient to a high risk of toxicity
13. A history of active autoimmune disease or possibly recurrent autoimmune disease that may affect vital organ function or require immunosuppressive therapy including systemic corticosteroids
14. Systemic treatment with either corticosteroid (> 10mg/ day prednisone) or other immunosuppressive drugs within 14 days of the study drug; Inhaled or topical steroids and adrenal-replacement doses (≤10mg per day of prednisone) were allowed in the absence of active autoimmune disease. Topical, intraocular, intra-articular, intranasal, and inhaled corticosteroids (with low systemic absorption) were allowed; Physiological alternative doses of systemic corticosteroids (≤10mg/ day prednisone) were allowed; Short-term corticosteroid therapy for prophylaxis (e.g., contrast allergy) or treatment of nonautoimmune conditions (e.g., delayed hypersensitivity due to contact allergens) was permitted
15. Bleeding tendency and history of thrombosis:

    1. Any bleeding event of CTCAE2 grade within 3 months before screening or of CTCAE grade 3 or higher within 6 months before screening
    2. They have active bleeding or abnormal coagulation function, have a tendency to bleed, or are receiving thrombolytic or anticoagulant therapy
    3. Patients require anticoagulant therapy with drugs such as warfarin or heparin
    4. Long-term antiplatelet therapy (e.g., aspirin, clopidogrel) is required.
    5. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism within the past 6 months
16. History of severe cardiovascular disease:

    1. New York Heart Association (NYHA) grade 3 and 4 congestive heart failure
    2. Unstable angina or newly diagnosed angina or myocardial infarction within 12 months before screening
    3. Arrhythmias requiring therapeutic intervention (patients taking beta-blockers or digoxin are eligible)
    4. CTCAE≥ grade 2 valvular heart disease
    5. Hypertension that cannot be controlled with medications (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg)
17. Patients who were pregnant or breastfeeding, or expected to plan to become pregnant during the study treatment
18. Any previous or current medical conditions, treatments, or laboratory abnormalities that may interfere with the results of the study or prevent the patient from participating fully in the study, or the investigator considers the patient to be unsuitable for the study; Patients could not receive platelet or red-cell transfusions for 4 weeks before starting the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 1 year
  Per RECIST v1.1 criteria, the proportion of patients whose best remission was CR or PR accounted for the total number of evaluable patients.

SECONDARY OUTCOMES:
Disease Control Rate | Time Frame: up to 1 year
  Per RECIST v1.1 criteria, the proportion of patients whose best remission was CR , PR and SD accounted for the total number of evaluable patients.
DOR | up to 2 years
  Duration of Response, determined according to RECIST v1.1 criteria
PFS | up to 2 years
  Progression Free Survival, determined according to RECIST v1.1 criteria
AEs | up to 1 years
  Adverse events defined according to Common Terminology for Adverse Events (CTCAE) v5.0
Overall survival（OS） | Up to 2 years
  Overall survival is the time from intervention to death due to any reason or lost of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided